CLINICAL TRIAL: NCT06215781
Title: Comparison Between Conventional and Digital Workflow in Fixed Dental Prosthetic Rehabilitations: a Randomized Clinical Trial Study
Brief Title: Comparison Between Conventional and Digital Workflow in Dental Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Massimo Corsalini, Prof, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UOC Odontostomatologia
Record Dates: First submitted 2023-12-27; First posted 2024-01-22 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Dental Prosthesis Complication

STUDY DESIGN:
Intervention Model Description: Three-arms groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fully digital workflow (Experimental): Patients of this group are subjected to entire digital workflow, from the digital planning to the delivery of definitive zirconia fixed dental prosthesis
  Interventions: Procedure: Fully digital workflow of prosthetic fixed dental crown
- Combined digital-conventional workflows (Experimental): Patients of this group were subjected to every digital steps as the "fully digital workflow" arm, except for the impression that includes analog material (silicones).
  Interventions: Procedure: Combined digital and conventional workflows of prosthetic fixed dental crown
- Fully conventional workflow (Active Comparator): Patients of this group follow the entire analog protocol. All the procedures exclude digital involvement.
  Interventions: Procedure: Fully conventional workflow of prosthetic fixed dental crown

INTERVENTIONS:
Procedure: Fully digital workflow of prosthetic fixed dental crown — The intervention that was administered was a full digital workflow. It includes an initial digital planning, an optical impression with intraoral scanner and a CAD-CAM milled zirconia crown. No analog materials were used.
  Arms: Fully digital workflow
Procedure: Combined digital and conventional workflows of prosthetic fixed dental crown — The intervention that was administered was a combined digital and traditional workflow. The initial planning was digital, then the impression was performed with analog impression material (silicones) and the final zirconia crown was CAD-CAM milled, with a digital procedure.
  Arms: Combined digital-conventional workflows
Procedure: Fully conventional workflow of prosthetic fixed dental crown — The intervention that was administered was a conventional workflow that doesn't provide any digital step. The impression was taken with analog material (silicones) and the final prosthesis was a metal-ceramic crown, realized on plaster cast.
  Arms: Fully conventional workflow

SUMMARY:
The aim of this comparative RCT is to evaluate the differences between the entire digital, the combined digital-analogic and the entire analogic workflows of implant-supported and teeth-supported prostheses. It is a three-arms comparative study. The 60 patients are divided into three groups:

* fully digital workflow
* combined digital and conventional workflow
* fully conventional workflow For each patients were evaluated the interproximal (IC) and occlusal contact (OC) and impression time (IT) and the patient satisfaction through a VAS scale.

The null hypothesis is that are no differences between the three groups for each parameter.

DETAILED DESCRIPTION:
This comparative RCT aims to evaluate the differences between the entire digital, the combined digital-analogic, and the entire analogic workflows of implant-supported and teeth-supported prostheses. It is a three-arms comparative study to better focus on the reliability of digital techniques.

Inclusion criteria were good oral health, absence of parafunction, no dental caries or presence of periodontitis, and healthy general conditions.

Exclusion criteria were bad oral health, parafunctions, dental caries or periodontitis, and general health comorbidities that don't allow surgical treatment.

The 60 patients are divided into three groups:

* fully digital workflow: each patient in this group was treated with an exclusively digital workflow, from digital planning of the surgical phase to digital impression and digital manufacturing of prosthetic crowns.
* combined digital and conventional workflow: each patient of this group was subjected to digital planning, and then, the impressions were taken with traditional analogical materials, so the plaster model was converted into a digital model, and there finally was performed a digital manufacturing of prosthetic crown.
* entirely conventional workflow: each patient was treated with an analogical technique. No digital phase was performed.

After prosthetic delivery, each patient were evaluated for interproximal (IC) and occlusal contact (OC), impression time (IT), and patient satisfaction through a VAS scale.

The null hypothesis is that there are no significant differences between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* good oral health
* good general health conditions
* no contraindication to oral surgery and fixed prosthesis
* patients who completed the 6 months follow-up

Exclusion Criteria:

* bad oral health
* bad general health conditions (with multi-drug therapy)
* periodontitis or dental caries susceptibly
* parafunctions presence
* TMJ disorders
* didn't accept the informed consent / treatment planning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Entity of interproximal contact | 2 weeks after definitive prosthesis delivery
  Precision of interproximal contact between prosthetic crown and adjacent teeth. It was measured by the clinician evaluating the resistance to the sliding of waxed dental floss. The clinician gives to the interproximal contact a score from 0 to 4, where 0 is considered as an absence of resistance (open space between crown and adjacent teeth) and 4 is the total impediment to the floss slide (the crown and the adjacent teeth are too close to have a correct interproximal contact)
Entity of occlusal contact | 2 weeks after definitive prosthesis delivery
  The entity of contact between prosthetic crown and antagonist teeth was evaluated with a dichromatic articulating paper in order to identify any static and dynamic alterations in occlusal contacts that must be corrected. The clinician gives a score from 0 to 3 where 0 is the absence of contact between crown and antagonists, 1 is a correct contact between them that needs no corrections, 2 there is a slight altered contact that requires minor corrections and 3 there is an altered contact between the prosthetic crown and their antagonists which requires major corrections.
Impression time | 2 weeks after definitive prosthesis delivery
  Length of time useful to take impression expressed in seconds
Patient satisfaction degree | 2 weeks after definitive prosthesis delivery
  Patient satisfaction through a VAS scale. The patients is asked to make a mark in an unnumbered line ranging from 0 to 5 where 0 represents maximum comfort and 5 represents a very bad experience. The scale is 5 cm long so the clinician next measures the distance (in cm) from 0 to where the mark was placed by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Corsalini, Prof., Principal Investigator — Interdisciplinary Department of Medicine, University of Bari "Aldo Moro"
Locations (1):
- Massimo Corsalini, Bari, Italy

IPD SHARING:
Plan to Share IPD: No
The database with study's outcomes will be shared on specific request.